CLINICAL TRIAL: NCT02721914
Title: The Effects of Massage Therapy and Hypopressive Abdominal Exercises on Chronic Non-specific Low Back Pain, Joint Mobility, Disability and the Patient's Quality of Life. A Controlled Clinical Trial
Brief Title: The Effectiveness of the Massage and the Hypopressive Abdominal Gymnastics on Low Back Pain (MAS-GAH)
Acronym: MAS-GAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Manuel Rebollo Salas, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USeville-MSalas
Record Dates: First submitted 2016-03-18; First posted 2016-03-29 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-01

CONDITIONS: Low-back Pain
Keywords: low-back pain; massage therapy; Gymnastics; disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- GROUP RECEIVING MASSOTHERAPY- HYPOPRESSIVE ABDOMINAL GYMNASTIC (Experimental): Subjects will receive 4 massotherapy sessions and 4 of HYPOPRESSIVE ABDOMINAL GYMNASTIC (HAG).
  Interventions: Procedure: GROUP RECEIVING MASSOTHERAPY- HYPOPRESSIVE ABDOMINAL GYMNASTIC
- GROUP RECEIVING MASSOTHERAPY (Experimental): The subjects of this group will receive a total of 8 sessions of 30 minutes each.
  Interventions: Procedure: GROUP RECEIVING MASSOTHERAPY
- GROUP RECEIVING HYPOPRESSIVE ABDOMINAL GYMNASTIC (Experimental): The subjects of this group will receive a total of 8 sessions of 30 minutes each.
  Interventions: Procedure: GROUP RECEIVING HYPOPRESSIVE ABDOMINAL GYMNASTIC

INTERVENTIONS:
Procedure: GROUP RECEIVING MASSOTHERAPY- HYPOPRESSIVE ABDOMINAL GYMNASTIC — The subjects of this group will receive an amount of eight sessions that will be applied within five weeks; four massotherapy sessions and another 4 of H.A.G. The three first weeks one session of each methodology will be applied, starting always with massotherapy (with sessions on Mondays and Thursdays or on Tuesdays and Fridays). On the fourth week a session of massotherapy will be applied on the same day as usual. And, finally, on the fifth week a session of H.A.G will be applied on the same day as massotherapy is applied.
  Arms: GROUP RECEIVING MASSOTHERAPY- HYPOPRESSIVE ABDOMINAL GYMNASTIC
Procedure: GROUP RECEIVING MASSOTHERAPY — The sessions will be applied for 5 weeks. The first three weeks 2 sessions per week will be applied (whether on Mondays and Thursdays or Tuesdays and Fridays), and during the remaining two weeks only a session will be applied per week, on the first day of the week same as applied before.
  Massotherapy technics will be applied all over the back, covering the thoracolumbar area as well as upper areas reaching the cervix and occiput.
  In particular, posterosuperior iliac spines, iliac crests, ribs, shoulder girdle and the entire spine (sacral bone- lumbar area-backbones-cervical vertebrae) and its attached tissues will be worked down.
  Massotherapy protocol will be applied by the physical therapist, always respecting the postural ergonomics. This enables the verticality of the body (avoiding the slopes) which makes work much easier thanks to the inertia triggered by the load transfer in the lower extremities in both sagittal and horizontal plane.
  Arms: GROUP RECEIVING MASSOTHERAPY
Procedure: GROUP RECEIVING HYPOPRESSIVE ABDOMINAL GYMNASTIC — The subjects of this group will receive a total of 8 sessions of 30 minutes each; sessions will be applied for 5 weeks. The first three weeks 2 sessions per week will be applied (whether on Mondays and Thursdays or Tuesdays and Fridays), and during the remaining two weeks only a session will be applied per week, on the first day of the week same as applied before.
  The techniques applied are an assembly of rhythm, postural and breathing exercises that have to be done in a systematically. The physical therapist will check that all of the group subjects have assimilated properly the H.A.G and the breathing patterns from the exercises protocol. If they have, then the practical session which comprises 6 hypopressive exercises, can be started.
  The subjects must remain in each position between 10 and 30 seconds and repeat the exercise three times, with a rest period among each that will last at least 20 seconds.
  Arms: GROUP RECEIVING HYPOPRESSIVE ABDOMINAL GYMNASTIC

SUMMARY:
The main goal of this study is to get to know if applying both, massotherapy plus hypopressive abdominal gymnastics (H.A.G) will reduce the pain of chronic non-specific low back pain. It actually reduces the inability produced by the pain and improve the patient's quality of life as well as the join range of the lumbar spine, way more than these two therapies applied separately.

DETAILED DESCRIPTION:
Background:

Back pain is one of the most common musculoskeletal disorders in the industrialized society. It is estimated to affect between 70 to 85% of the adult population over their live. The impact of low back pain is widespread in developed countries, and accounts the major spending in economic and health resources, as well as being associated with the leading causes of absenteeism and disability. Diagnosis, in most cases, nonspecific low back pain, the symptoms have no clear cause, so that the source of pain is unknown. In general, a significant percentage progresses to chronic back pain and is accompanied by a limitation of physical activity influenced by improper posture or movement patterns.

Objectives:

To assess the effectiveness of massage therapy and hypopressive abdominal gymnastics, and the combination of both therapeutic modalities, to decrease pain and lumbar disability; and increasing joint mobility and quality of life in patients with chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic non-specific low back pain diagnosed and at least 12 weeks of mechanical pain.

Exclusion Criteria:

* Patients:
* With arterial hypertension diagnosed.
* With progressive neurological deficits.
* Pregnant or suspect that they are pregnant.
* With psychological or psychiatric process diagnosed.
* Under analgesic treatment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from Self-reported lumbar pain intensity at 3 weeks. | At the start of the study, before the fifth treatment session (third week)
  Evaluated by the numerical pain scale.
Change from Self-reported lumbar pain intensity at 5 weeks. | After the last treatment session (fifth week).
  Measured by the Oswestry disability index.
Change from Disability at 3 weeks. | At the start of the study, before the fifth treatment session (third week)
  Measured by the Oswestry disability index.
Change from Disability at 5 weeks. | After the last treatment session (fifth week).
  Measured by the Oswestry disability index.

SECONDARY OUTCOMES:
Change from Lumbar joint mobility at 3 weeks. | At the start of the study, before the fifth treatment session (third week)
  Lumbar flexion measured by the modified Schober test
Change from Lumbar joint mobility at 5 weeks. | After the last treatment session (fifth week).
  Lumbar flexion measured by the modified Schober test
Change from Quality of life at 3 weeks. | At the start of the study, before the fifth treatment session (third week)
  Measured by the Short-Form-12 Health Survey
Change from Quality of life at 5 weeks. | After the last treatment session (fifth week).
  Measured by the Short-Form-12 Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Seville, Spain

REFERENCES:
- [Background] Trampas A, Mpeneka A, Malliou V, Godolias G, Vlachakis P. Immediate Effects of Core-Stability Exercises and Clinical Massage on Dynamic-Balance Performance of Patients With Chronic Specific Low Back Pain. J Sport Rehabil. 2015 Nov;24(4):373-83. doi: 10.1123/jsr.2014-0215. Epub 2014 Dec 4. PMID 25474502
- [Result] Resende AP, Torelli L, Zanetti MR, Petricelli CD, Jarmy-Di Bella ZI, Nakamura MU, Araujo Junior E, Moron AF, Girao MJ, Sartori MG. Can Abdominal Hypopressive Technique Change Levator Hiatus Area?: A 3-Dimensional Ultrasound Study. Ultrasound Q. 2016 Jun;32(2):175-9. doi: 10.1097/RUQ.0000000000000181. PMID 26441380
- [Result] Stupp L, Resende AP, Petricelli CD, Nakamura MU, Alexandre SM, Zanetti MR. Pelvic floor muscle and transversus abdominis activation in abdominal hypopressive technique through surface electromyography. Neurourol Urodyn. 2011 Nov;30(8):1518-21. doi: 10.1002/nau.21151. Epub 2011 Aug 8. PMID 21826719
- [Result] Chou R, Deyo R, Friedly J, Skelly A, Hashimoto R, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S, Brodt E. Noninvasive Treatments for Low Back Pain [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2016 Feb. Report No.: 16-EHC004-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK350276/ PMID 26985522
- [Result] Sejari N, Kamaruddin K, Ramasamy K, Lim SM, Neoh CF, Ming LC. The immediate effect of traditional Malay massage on substance P, inflammatory mediators, pain scale and functional outcome among patients with low back pain: study protocol of a randomised controlled trial. BMC Complement Altern Med. 2016 Jan 15;16:16. doi: 10.1186/s12906-016-0988-1. PMID 26767971
- [Result] Furlan AD, Giraldo M, Baskwill A, Irvin E, Imamura M. Massage for low-back pain. Cochrane Database Syst Rev. 2015 Sep 1;2015(9):CD001929. doi: 10.1002/14651858.CD001929.pub3. PMID 26329399
- [Derived] Bellido-Fernandez L, Jimenez-Rejano JJ, Chillon-Martinez R, Lorenzo-Munoz A, Pinero-Pinto E, Rebollo-Salas M. Clinical relevance of massage therapy and abdominal hypopressive gymnastics on chronic nonspecific low back pain: a randomized controlled trial. Disabil Rehabil. 2022 Aug;44(16):4233-4240. doi: 10.1080/09638288.2021.1884903. Epub 2021 Feb 15. PMID 33587856
- [Derived] Bellido-Fernandez L, Jimenez-Rejano JJ, Chillon-Martinez R, Gomez-Benitez MA, De-La-Casa-Almeida M, Rebollo-Salas M. Effectiveness of Massage Therapy and Abdominal Hypopressive Gymnastics in Nonspecific Chronic Low Back Pain: A Randomized Controlled Pilot Study. Evid Based Complement Alternat Med. 2018 Feb 22;2018:3684194. doi: 10.1155/2018/3684194. eCollection 2018. PMID 29681973